CLINICAL TRIAL: NCT06721065
Title: RSMI HEALS (Health Equity Advances Through Language Solutions) (AI)
Brief Title: A Study of Language Interpretation Solutions for People With Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-350
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Breast Cancer Stage II; Breast Cancer Stage III
Keywords: Breast Cancer; Breast Cancer Stage II; Breast Cancer Stage III; Language Interpretation; Spanish; Mandarin; Memorial Sloan Kettering Cancer Center; 24-350
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase I: Remote Simultaneous Medical Interpreting/RSMI (Arm 1) (Experimental): This phase will enroll Spanish- and Mandarin-speaking patients with LEP (Stages II and III disease) and English- speaking providers
  Interventions: Other: Remote Simultaneous Medical Interpreting/RSMI
- Phase I: Remote Consecutive Medical Interpreting/RCMI (Arm 2) (Experimental): This phase will enroll Spanish- and Mandarin-speaking patients with LEP (Stages II and III disease) and English- speaking providers
  Interventions: Other: Remote Consecutive Medical Interpreting/RCMI
- Phase I: Remote Consecutive Video Medical Interpreting/RCVI (Arm 3) (Experimental): This phase will enroll Spanish- and Mandarin-speaking patients with LEP (Stages II and III disease) and English- speaking providers
  Interventions: Other: Remote Consecutive Video Medical Interpreting/RCVI
- Phase II: CFIR mixed-methods explanatory, multi- stakeholder process evaluation (Experimental): Will examine RSMI utilization (Arm 1 participants only and clinic staff), intervention barriers and facilitators, and implementation potential
  Interventions: Other: Remote Simultaneous Medical Interpreting/RSMI

INTERVENTIONS:
Other: Remote Simultaneous Medical Interpreting/RSMI — Remote Simultaneous Medical Interpreting (RSMI), "UN-style" simultaneous interpreting applied to the medical encounter, which holds tremendous promise for closely approximating a same language encounter, decreasing interpreting errors, and improving outcomes.
  Arms: Phase I: Remote Simultaneous Medical Interpreting/RSMI (Arm 1); Phase II: CFIR mixed-methods explanatory, multi- stakeholder process evaluation
Other: Remote Consecutive Medical Interpreting/RCMI — Remote Consecutive Medical Interpreting (RCMI; "audio consecutive"), is the most commonly utilized remote interpreting
  Arms: Phase I: Remote Consecutive Medical Interpreting/RCMI (Arm 2)
Other: Remote Consecutive Video Medical Interpreting/RCVI — Remote Simultaneous Medical Interpreting (RSMI), "UN-style" simultaneous interpreting applied to the medical encounter
  Arms: Phase I: Remote Consecutive Video Medical Interpreting/RCVI (Arm 3)

SUMMARY:
The study will be conducted in 2 overlapping phases. In Phase 1, there will be a 3-arm randomized controlled trial of Remote Simultaneous Medical Interpreting/RSMI (Arm 1), versus Remote Consecutive Medical Interpreting/RCMI (Arm 2) and versus Remote Consecutive Video Medical Interpreting/RCVI (Arm 3) in breast cancer outpatient clinical encounters with Spanish- and Mandarin-speaking patients with Limited English Proficiency/LEP (Stages II and III disease) and English- speaking providers (who do not speak Spanish/Mandarin). In Phase 2, there will be a sequential mixed-methods explanatory, multi-stakeholder process evaluation to gather implementation potential data.

ELIGIBILITY:
Inclusion Criteria:

Phase I Patients

* Age >=18 years (per EMR)
* Preferred language for healthcare is Spanish or Mandarin (per self-report)
* Limited English Proficient; cannot speak English "very well" (per self-report)
* Diagnosis of breast cancer or gastrointestinal (per EMR)
* Will be visiting MSK oncology teams for the first or second appointment (per EMR)
* Agrees to be audio-recorded (per self-report)

Phase 1 Providers

* Breast or gastrointestinal cancer provider who sees patients (e.g., breast or gastrointestinal oncologists, advanced practice providers, and/or nurses)
* Does not speak Spanish and/or Mandarin; providers who speak one language and not the other may participate (e.g., speaks Spanish but not Mandarin) (per self-report)
* Agrees to be audio-record (per self-report) Phase 2 (clinic staff only; patient participants will be drawn from Phase 1)
* Is a staff member who works/worked in one of the study clinic sites during the period of Phase 1 RCT study activities
* Agrees to be audio-recorded (per self-report)

Exclusion Criteria:

Phase 1 Patients

* Has significant psychiatric disturbance (i.e., acute psychiatric symptoms) sufficient to preclude completion of the assessments, interviews, or informed consent (per EMR, patient's care team, or study team)
* Presence of cognitive impairment disorder (i.e., delirium or dementia) sufficient to preclude meaningful informed consent and/or data collection (per EMR, patients, care team, or study team)

Phase I Providers

* None

Phase 2 (clinic staff only; Phase 1 patient participants follow above criteria)

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2029-12-02 (Estimated); Study Completion 2029-12-02 (Estimated)

PRIMARY OUTCOMES:
Number of interpretation errors | up to 30 days
  Via translation and transcription of audio recordings, errors will be determined in the interpretation of medical facts made in each of the RCT arms during Study Visit 1 (post- diagnosis)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Gany, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk- Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent Only), Harrison, New York
  - Memorial Sloan Kettering at Ralph Lauren Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org